CLINICAL TRIAL: NCT03272581
Title: The Effects of Functional Training on Performance Related Physical Fitness Parameters in Professional Basketball Players
Brief Title: The Purpose of This Study Was to Determine Whether or Not Functional Training Has Similar Effects on Muscular Strength, Flexibility, Agility, Speed and Anthropometric Measures in Basketball Players as Traditional Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Serkan Usgu, Assistant Professor of Physiotherapy and Rehabilitation, Hasan Kalyoncu University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUT 12/99-24
Record Dates: First submitted 2017-08-25; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Basketball; Exercise
Keywords: Functional; Training; Performance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Control group followed routine basketball training and traditional strength training.
- Training Group (Experimental): Functional exercises were applied to training group for 20 weeks (2 days/week) with routine basketball training.
  Interventions: Other: Functional Training

INTERVENTIONS:
Other: Functional Training — Functional training has been defined as emphasizing multiple muscle and joint activities, combining upper and lower body movements, and utilizing more of the body in each movement. The primary goal of functional training is to transfer improvement achieve in one movement to enhancing the performance of another movement by affecting the entire neuromuscular system.
  Arms: Training Group

SUMMARY:
Basketball has gained worldwide popularity and fascinated players and spectators with its dynamic characteristics as a team sport. This kind of sport is multifaceted that requires well-developed physical ﬁtness to be played successfully. Many authors have suggested that strength, power, agility, and speed are important performance related physical components for elite basketball players. The physical components require that fitness and conditioning attributes of basketball players are well developed to negate the limiting aspect of sport performance. Moreover, functional training is becoming increasingly popular within the fitness industry and has been considered to be a better alternative than traditional training methods for improving various measures of performance. The purpose of this study was to determine whether functional training has effects on performance and related various physical components of basketball players.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be professional basketball players
* Participants have not any upper or lower extremities injury during last 3 months
* Participants must implement age limits

Exclusion Criteria:

* If participants who has;

  1. Surgery
  2. Musculoskeletal injuries
* Participants who transfer to another professional basketball team
* If participants who has;

  1. Systematic inflammatory diseases
  2. Neurological diseases
  3. Vascular conditions
  4. Alcohol abuse
  5. Psychiatric disorders

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2014-01-29 (Actual); Study Completion 2015-03-17 (Actual)

PRIMARY OUTCOMES:
one repetition strength tests | 20 weeks
  maximal bench press and leg press tests
jump tests | 20 weeks
  standing broad jump and vertical jump

SECONDARY OUTCOMES:
Speed Test | 20 weeks
  20 meters speed test
Agility tests | 20 weeks
  T-Drill and Lane-Agility tests
Flexibility Test | 20 weeks
  Sit and reach test

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Usgu, PhD, Principal Investigator — Hasan Kalyoncu University; Günseli Usgu, PhD, Principal Investigator — Hasan Kalyoncu University; Yavuz Yakut, Prof, Principal Investigator — Hasan Kalyoncu University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code

REFERENCES:
- [Result] Lagally KM, Cordero J, Good J, Brown DD, McCaw ST. Physiologic and metabolic responses to a continuous functional resistance exercise workout. J Strength Cond Res. 2009 Mar;23(2):373-9. doi: 10.1519/JSC.0b013e31818eb1c9. PMID 19197213
- [Result] Boyle, M., Functional training for sports. 2004: Human Kinetics
- [Result] Whitehurst MA, Johnson BL, Parker CM, Brown LE, Ford AM. The benefits of a functional exercise circuit for older adults. J Strength Cond Res. 2005 Aug;19(3):647-51. doi: 10.1519/R-14964.1. PMID 16095420
- [Result] de Vreede PL, Samson MM, van Meeteren NL, Duursma SA, Verhaar HJ. Functional-task exercise versus resistance strength exercise to improve daily function in older women: a randomized, controlled trial. J Am Geriatr Soc. 2005 Jan;53(1):2-10. doi: 10.1111/j.1532-5415.2005.53003.x. PMID 15667369
- [Result] Kibele A, Behm DG. Seven weeks of instability and traditional resistance training effects on strength, balance and functional performance. J Strength Cond Res. 2009 Dec;23(9):2443-50. doi: 10.1519/JSC.0b013e3181bf0489. PMID 19952576
- [Result] Milton, D.E., et al., The effect of functional exercise training on functional fitness levels of older adults. 2006, University of Wisconsin--La Crosse.
- [Result] Weiss, T., et al., Effect of functional resistance training on muscular fitness outcomes in young adults. Journal of Exercise Science & Fitness, 2010. 8(2): p. 113-122
- [Result] Oliver GD, Di Brezzo R. Functional balance training in collegiate women athletes. J Strength Cond Res. 2009 Oct;23(7):2124-9. doi: 10.1519/JSC.0b013e3181b3dd9e. PMID 19855341
- [Result] Thompson CJ, Cobb KM, Blackwell J. Functional training improves club head speed and functional fitness in older golfers. J Strength Cond Res. 2007 Feb;21(1):131-7. doi: 10.1519/00124278-200702000-00024. PMID 17313268
- [Result] Murugan, A., Nageswaran, A. (2014) İnfluence of functional training on selected physical components among cricketers. Journal of Recent Research and Applied Studies, 1 (2(5)).
- [Result] Myer GD, Ford KR, Palumbo JP, Hewett TE. Neuromuscular training improves performance and lower-extremity biomechanics in female athletes. J Strength Cond Res. 2005 Feb;19(1):51-60. doi: 10.1519/13643.1. PMID 15705045